CLINICAL TRIAL: NCT06765811
Title: Identification of Rapid Kidney Function Decline in Older Adults with Different Types of Aging
Brief Title: Rapid Kidney Function Decline in Older Adults
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Professor, Huashan Hospital
Other Study IDs: KY2024-1068
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-07

CONDITIONS: Kidney Function Decline; Glomerular Filtration Rate; Urine Albumin-creatinine Ratio; Healthy Aging; Comorbidity; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rugao Longevity and Aging Study (RLAS) cohort: A total of 1,236 older adults from the Rugao Longevity and Aging Study (RLAS) were enrolled in the study, including 575 healthy aging individuals and 661 with comorbid co-morbidities (e.g., diabetes mellitus, hypertension, coronary heart disease, etc.). The objective of the study was twofold: first, to assess the predictive value of baseline glomerular filtration rate (GFR) to urinary albumin-creatinine ratio (ACR) for rapid decline in renal function (≥30% decline in GFR) within 2 years; and second, to establish early warning criteria for different types of aging populations.
- Healthcare data from Huashan Hospital, Fudan University (CKD): The present cohort comprised 303 elderly patients suffering from chronic kidney disease (CKD) from Huashan Hospital of Fudan University, including cases progressing from acute kidney injury (AKI) to CKD. The objective of the study was twofold: first, to assess the predictive ability of baseline GFR and ACR levels for rapid decline in renal function (≥30% GFR) within two years; and second, to establish appropriate early risk assessment criteria for the elderly CKD population.

SUMMARY:
This observational study investigates whether a single set of GFR and urine albumin-to-creatinine ratio (ACR) thresholds can accurately screen for rapid kidney function decline in different elderly groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 70 years;
2. GFR data measured at least twice (two years apart) and ACR data measured once (at baseline);
3. A clear record of the cause of the previous visit; from this, people diagnosed with kidney disease were selected, and kidney disease was defined as various primary nephritis, secondary nephropathy, acute kidney injury (AKI), chronic kidney disease, kidney tumors, or a diagnosis of proteinuria alone.
4. Signed informed consent form.

Exclusion Criteria:

1. People with missing baseline biochemical data;
2. Outliers in the population indicators, i.e., data deviating from the mean ± three times the standard deviation;
3. Data with significantly abnormal baseline renal function follow-up (abnormally elevated GFR by more than 10% within 2 years or abnormal ACR value as determined by consultation with a senior nephrologist).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: kidney disease patient
Sampling Method: Non-Probability Sample
Enrollment: 1539 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
A ≥30% decline in glomerular filtration rate (GFR) within 2 years, i.e. a rapid decline in renal function | The risk of rapid decline in kidney function in the elderly was assessed during a 2-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital, Fudan university, Shanghai, Shanghai Municipality, China